CLINICAL TRIAL: NCT01105520
Title: Neurologic and Neurophysiologic Assessment of Clinical Course in Patients With Intraspinal Processes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Prof. H. Bertalanffy, University of Zurich
Other Study IDs: ZU-XYZ-003
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Tumor
Keywords: Intraspinal processes (tumor or vascular malformation AVM)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- intralspinal processes: Patients with intralspinal processes
  Interventions: Procedure: Diagnostic

INTERVENTIONS:
Procedure: Diagnostic — SCIM Spinal Cord Independence Measure ASIA scale American Spinal Injury Association

SUMMARY:
Patients included in the study are treated at the Klinik für Neurochirurgie USZ. The clinical course is documented at Paraplegikerzentrum Balgrist using validated diagnostic procedures (e.g. SCIM, ASIA, neurophysiology).

Study aims:

Prognostic value of clinical diagnosis and additional diagnostic procedures? Which parameters exhibit optimal prognostic power? Differences between tumor/AVM associated lesions and traumatic lesions? What can we learn for pathophysiology and treatment?

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* Benign intraspinal process (tumor or vascular malformation AVM)
* Primary lesion caudal of the brainstem, affecting C1
* Cognitive ability to give written informed consent

Exclusion criteria:

* Metastases, malign tumors
* Traumatic lesions
* Myelitis, polyneuropathy
* Disc prolaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated surgically for intraspinal processes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Study Completion 2015-12

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland